CLINICAL TRIAL: NCT03392688
Title: Is There a Time Difference Between Onsets of Lateral and Medial Hamstring Muscles During Gait in Patients With Patellofemoral Pain Comparing to Healthy Subjects?
Brief Title: Time Difference Between Onsets of Lateral And Medial Hamstring Muscles During Gait in Patients With Patellofemoral Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Dilber Karagozoglu Coskunsu, Assistant Professor, Bahçeşehir University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: BahcesehirU
Record Dates: First submitted 2017-12-20; First posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Patellofemoral Pain
Keywords: onset , hamstring muscles, patellofemoral pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Electromyography

STUDY DESIGN:
Intervention Model Description: Participants which were included in the study were divided into 2 groups as patient group who included the patients diagnosed with Patellofemoral pain and asymptomatic group which was considered as control group.
Who Masked: Outcomes Assessor
Masking Description: The algorithm used to calculate the onset of the EMG was identified according to the point at which the signal deviated by more than three times standard deviations, for a minimum of 25 ms from the baseline level (computing started 200 ms prior to the start of walking). MatLab program (R2011 version) was used for design a custom made program for data analysis. Additionally to automatic calculation, all data was visually checked to ensure that there was no signal noise, deteriorating the signal analysis, possibly caused by the movement artefact. A blind assessor visualy checked the onsets of the MH and LH muscles and record the onset time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patellofemoral pain group (Experimental): Diagnosis of PFP was established based on symptoms, physical examination performed by an orthopedic surgeon. Patients were also screened through physical examination to rule out ligamentous or meniscal injuries, patellar tendinitis and knee joint effusion by an orthopedic surgeon. All patients also underwent a radiologic examination consisting of AP, lateral and tangential radiograms.
  Surface EMG, Kujala patellofemoral pain scale, Q angle measurement were administered to the PFP group.
  Interventions: Other: kujala patellofemoral pain scale; Diagnostic Test: Surface EMG; Other: Q angle measurement
- Control Group (Active Comparator): Control group had similar demographic characteristics with PFP group, and neither one of the controls had any knee pathology or current knee pain or effusion that would effect the gait.
  Surface EMG, Q angle measurement were administered to the control group.
  Interventions: Diagnostic Test: Surface EMG; Other: Q angle measurement

INTERVENTIONS:
Other: kujala patellofemoral pain scale — Kujala patellofemoral pain scale was used to evaluate knee functions of the PFP subjects.
  Arms: Patellofemoral pain group
Diagnostic Test: Surface EMG — The surface EMG electrodes (silver/silver chloride, pre-gelled, Ambu Blue Sensor, Denmark) (Konrad P.) with an interelectrode distance of 20 mm between centers were used to record an EMG signal during walking. Portable 8 channel (TELEEMG, BTS, Milan, Italy) with built in x10 amplifications, 10-450 Hz bandpass and sampling rate of 1000 Hz were used for recording. The location and orientation of the electrodes for each MH (ST) and LH (BF) were identified according to SENIAM (Surface ElectromyoGraphy for the Non-Invasive Assessment of Muscles) criteria.
Other: Q angle measurement — Q angle measurement was applied to both patellofemoral pain and control group subjects in standing position.

SUMMARY:
Early activation of lateral hamstrings (LH) in respect of medial hamstrings (MH) may cause abnormal knee abduction and external rotation moments in individuals. This situation may increase the risk of ligament injury and may be the reason for susceptibility of patellofemoral pain (PFP). The aim of this study is to compare the time delays in electromyographic studies between medial and lateral hamstrings in patients with PFP and asymptomatic subjects.

DETAILED DESCRIPTION:
Patellofemoral pain (PFP) is a very common complaint in younger population with still unclear and controversial etiology. It was suggested that a combination of intrinsic and extrinsic factors cause PFP. The strain of the retropatellar subcondral bone caused by excessive lateral patellar tracking is known to be the one among intrinsic factors (Thomee R.1999). Imbalance of the dynamics between knee extensor muscles, Vastus Medialis (VM) and Vastus Lateralis (VL), has also received a great research interest during last 10 years. However, uneven timing between onsets of counterpart knee flexor muscles, Lateral and Medial hamstring, were just considered as a possible etiological factor of the PFP (Patil S.2011), yet this hypothesis remains to be proven. The investigators aimed to investigate whether there is a relative time delays of the LH (biceps femoris, BF) and MH (semitendinosus, ST) during the walking at the self-selected speed in patients with patellofemoral pain. Even though dynamic EMG investigations are challenging because of cross-talks between muscles, hence difficult to determine clearly onset times, the investigators think that any information acquired during walking would be highly important because patellofemoral pain is mainly exaggerated by dynamic activities.

15 patients who were diagnosed with PFP (age 28.73±7.44, height 169.73±7.09, weight 67.47±14.31) and 15 asymptomatic subjects (age 30.47±6.22, height 167.87±7.81, weight 67.87±13.48) were recruited in the study. The inclusion criteria for PFP subjects was presence of the anterior and retropatellar pain for minimum 2 months scaled as 3 in accordance with Numeric Analog Scale during at least two of the following activities: stair descending, ascending, squatting, prolonged sitting, jumping, sitting on the knees. Surface EMG was recorded from Medial Hamstring and Lateral Hamstring muscles at 1000 Hz sampling rate during walking at participants' normal walking speed. EMG data obtained from 5 gait trials were evaluated. The EMG traces were full wave rectified and low pass filtered at 50 Hz. Delay in timing before heel strikes between MH and LH was calculated. Statistical significance between differences in time delays was analysed using "paired sample t-test".

ELIGIBILITY:
Inclusion Criterias:

* Pain originating specifically from the patellofemoral articulation (vague or localized);
* At least 3/10 pain intensity accordingly to the Numeric Analog Scale (NAS) with at least 2 of the following functional activities commonly associated with PFP stair ascent or descent, squatting, kneeling, or prolonged sitting;
* Reports of pain greater than 2 months in duration.
* Being between 18-40 years of age

Exclusion Criterias:

* Previous history of knee surgery,
* History of patellar instability,
* Neurologic involvement that would influence gait

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01-21 (Actual); Primary Completion 2015-05-30 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
Time difference between the onsets of the medial and lateral hamstring muscles | Preparing participants that include skin preparation and electrodes placement, and recording EMG data took average one hour for each participant
  The surface EMG electrodes (silver/silver chloride, pre-gelled, Ambu Blue Sensor, Denmark) (Konrad P.) with an interelectrode distance of 20 mm between centers were used to record an EMG signal during walking. Portable 8 channel (TELEEMG, BTS, Milan, Italy) with built in x10 amplifications, 10-450 Hz bandpass and sampling rate of 1000 Hz were used for recording. The location and orientation of the electrodes for each MH (ST) and LH (BF) were identified according to SENIAM (Surface ElectromyoGraphy for the Non-Invasive Assessment of Muscles) criteria

SECONDARY OUTCOMES:
kujala patellofemoral pain scale | At the begining of the study each participant was asked to complete the scale. It took average 10 minutes. Performed once.
  Kujala patellofemoral pain scale (Kujala 1993) is composed of 13 items that evaluate subjective symptoms and functional limitations. Minimum score is 0 points and maximum score is 100 points; higher values represent a worse outcome. Kujala patellofemoral pain scale is reported to be responsive, valid and demonstrates high test-retest reliability (Crosley K.2014). Turkish version of the Kujala patellofemoral pain score was used in our study (Kuru T. 2010).
Numeric Rating Scale (NRS) | Performed 1 day once.
  The NRS is an 11-point scale consisting of integers from 0 through 10; 0 representing ''No pain'' and 10 representing ''Worst imaginable pain.'' Participants select the single number that best represents their pain intensity.
Q angle | Performed 1 day once.
  Q angle measurement in standing

CONTACTS AND LOCATIONS:
Overall Officials: Dilber Karagozoglu Coskunsu, Ass. Prof., Principal Investigator — Bahcesehir University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation; Filiz Can, Prof., Study Director — Hacettepe University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation; Necla Ozturk, Prof., Study Chair — Maltepe University, Faculty of Medicine, Deparment of Biophysics; N. Ekin Akalın, Prof., Study Chair — Kultur University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation
Locations (1):
- Istanbul University,Faculty of Medicine, Deparment of Orthopedics and Traumatology, Gait Analysis Laboratory, Istanbul, Europe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication

REFERENCES:
- [Background] Patil S, Dixon J, White LC, Jones AP, Hui AC. An electromyographic exploratory study comparing the difference in the onset of hamstring and quadriceps contraction in patients with anterior knee pain. Knee. 2011 Oct;18(5):329-32. doi: 10.1016/j.knee.2010.07.007. Epub 2010 Aug 17. PMID 20724165
- [Background] Cowan S.M , Bennell K.L., Hodges P.W, Mc Connel J (2000). The test-retest reliability of the onset of concentric and eccentric vastus medialis obliquus and vastus lateralis electromyographic activity in a stair stepping task. Physical Therapy in Sport. 1, 129-136.
- [Background] Ng EC, Chui MP, Siu AY, Yam VW, Ng GY. Ankle positioning and knee perturbation affect temporal recruitment of the vasti muscles in people with patellofemoral pain. Physiotherapy. 2011 Mar;97(1):65-70. doi: 10.1016/j.physio.2010.05.009. PMID 21295240
- [Background] Li G, DeFrate LE, Zayontz S, Park SE, Gill TJ. The effect of tibiofemoral joint kinematics on patellofemoral contact pressures under simulated muscle loads. J Orthop Res. 2004 Jul;22(4):801-6. doi: 10.1016/j.orthres.2003.11.011. PMID 15183437